CLINICAL TRIAL: NCT04880655
Title: A Randomized, Controlled Study Evaluating a Surfactant-based Wound Dressing for Tissue Salvage and Reduction in Surgical Burden
Brief Title: A Randomized Trial Evaluating EARLY Application of a Surfactant Dressing in Thermal Injury (EARLY)
Acronym: EARLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-07861-XP
Record Dates: First submitted 2021-05-03; First posted 2021-05-11 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Burns; Partial-thickness Burn
Keywords: EARLY; Randomized Clinical Trial; Surfactant; Dressing; Total Body Surface Area; Outcome Assessment; Thermal Burn Injuries
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention (Experimental): Dressed with WSD and petrolatum gauze
  Interventions: Device: WSD
- Control (Active Comparator): Dressed with bacitracin and petrolatum gauze
  Interventions: Device: Dressed with bacitracin and petrolatum gauze

INTERVENTIONS:
Device: WSD — Post debridement and within 24 hours of injury, wound care and WSD applied daily
  Arms: Intervention
Device: Dressed with bacitracin and petrolatum gauze — Post debridement and within 24 hours of injury, wound care and dressing applied daily
  Arms: Control

SUMMARY:
The purpose of this study is to test the following hypotheses:

1. Early use of water-soluble surfactant dressing (WSD) on partial-thickness burn wounds will result in tissue salvage and reduce surgical burden.
2. Early use of WSD on partial-thickness burn wounds will result in faster healing.
3. Use of WSD on partial-thickness burn wounds will result in less painful wound care.
4. Early use of WSD on partial-thickness burn wounds will result in less infection.
5. Early use of WSD on partial-thickness burn wounds will result in lower hospital costs.

DETAILED DESCRIPTION:
Surfactant-based wound dressings have been utilized in chronic, non-healing wounds and small burn wounds to soften and aid removal of wound debris. In vitro data suggest enhanced healing properties are due the ability to stabilize and potentially reseal plasma membranes, thereby, retaining cellular integrity and enhance wound healing. Improved cellular viability and functionality has also been established in heat-shock, ionizing radiation, and electrical injury models. In one rat model, topically suffused mesentery demonstrated improved microvascular flow and reduction in the number of abnormally flowing microvessels following thermal injury. Intravenous administration has been studied in several disease states. In thermal injury, intravenous administration has shown potential to improve blood flow and reduce the zone of coagulation. Further, surfactant-based wound dressings are non-ionic and may facilitate removal, sensitize, or prevent bacterial biofilms. Biofilms are an evolved, protective mechanism bacteria utilize to reduce antimicrobial efficacy. Removal or penetration of biofilms is essential for bacterial eradication. There is little evidence demonstrating the efficacy of early use of a WSD for treating partial-thickness burn wounds.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* admitted within 24 hours of injury
* partial-thickness burn wounds on at least two non-contiguous areas of < 10% TBSA each and not involving face, fingers, toes, and perineum
* initial management assessed to require inpatient care

Exclusion Criteria:

* chemical, electrical, or inhalation injury
* pregnant
* incarcerated
* TBSA ≥ 20%
* wound expected to heal within 7 days
* patient or authorized representative unable or unwilling to consent
* unable to consent within 24 hours of injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Percent difference (cm2) in partial-thickness wound conversion | Up to 14 days
  Tissue salvage

SECONDARY OUTCOMES:
Time to 95% re-epithelialization | Up to 28 days
  Healing time
Daily pain scores for each wound care session | Up to 7 days
  Pain via Numeric Rating Scale (0-10; 0 having no pain and 10 being the worst possible pain)
Incidence of burn wound infection and cellulitis | Up to 28 days
  Infection up to day of initial excision or day of discharge
Hospital costs | Up to 28 days
  Cost of care during inpatient stay

CONTACTS AND LOCATIONS:
Locations (1):
- Regional One Health, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palumbo FP, Harding KG, Abbritti F, Bradbury S, Cech JD, Ivins N, Klein D, Menzinger G, Meuleneire F, Seratoni S, Zolss C, Mayer D. New Surfactant-based Dressing Product to Improve Wound Closure Rates of Nonhealing Wounds: A European Multicenter Study Including 1036 Patients. Wounds. 2016 Jul;28(7):233-40. PMID 27428718
- [Background] Birchenough SA, Rodeheaver GT, Morgan RF, Peirce SM, Katz AJ. Topical poloxamer-188 improves blood flow following thermal injury in rat mesenteric microvasculature. Ann Plast Surg. 2008 May;60(5):584-8. doi: 10.1097/SAP.0b013e3181651661. PMID 18434836
- [Background] Rodeheaver GT, Kurtz L, Kircher BJ, Edlich RF. Pluronic F-68: a promising new skin wound cleanser. Ann Emerg Med. 1980 Nov;9(11):572-6. doi: 10.1016/s0196-0644(80)80228-9. PMID 7436067
- [Background] Chen R, Salisbury AM, Percival SL. In vitro cellular viability studies on a concentrated surfactant-based wound dressing. Int Wound J. 2019 Jun;16(3):703-712. doi: 10.1111/iwj.13084. Epub 2019 Mar 20. PMID 30895731
- [Background] Maskarinec SA, Wu G, Lee KY. Membrane sealing by polymers. Ann N Y Acad Sci. 2005 Dec;1066:310-20. doi: 10.1196/annals.1363.018. PMID 16533934
- [Background] Lee RC, Hannig J, Matthews KL, Myerov A, Chen CT. Pharmaceutical therapies for sealing of permeabilized cell membranes in electrical injuries. Ann N Y Acad Sci. 1999 Oct 30;888:266-73. doi: 10.1111/j.1749-6632.1999.tb07961.x. PMID 10842638
- [Background] Lee RC, River LP, Pan FS, Ji L, Wollmann RL. Surfactant-induced sealing of electropermeabilized skeletal muscle membranes in vivo. Proc Natl Acad Sci U S A. 1992 May 15;89(10):4524-8. doi: 10.1073/pnas.89.10.4524. PMID 1584787
- [Background] Walsh AM, Mustafi D, Makinen MW, Lee RC. A surfactant copolymer facilitates functional recovery of heat-denatured lysozyme. Ann N Y Acad Sci. 2005 Dec;1066:321-7. doi: 10.1196/annals.1363.029. PMID 16533935
- [Background] Greenebaum B, Blossfield K, Hannig J, Carrillo CS, Beckett MA, Weichselbaum RR, Lee RC. Poloxamer 188 prevents acute necrosis of adult skeletal muscle cells following high-dose irradiation. Burns. 2004 Sep;30(6):539-47. doi: 10.1016/j.burns.2004.02.009. PMID 15302418
- [Background] Baskaran H, Toner M, Yarmush ML, Berthiaume F. Poloxamer-188 improves capillary blood flow and tissue viability in a cutaneous burn wound. J Surg Res. 2001 Nov;101(1):56-61. doi: 10.1006/jsre.2001.6262. PMID 11676555
- [Background] Yang Q, Schultz GS, Gibson DJ. A Surfactant-Based Dressing to Treat and Prevent Acinetobacter baumannii Biofilms. J Burn Care Res. 2018 Aug 17;39(5):766-770. doi: 10.1093/jbcr/irx041. PMID 29931339
- [Background] Yang Q, Larose C, Della Porta AC, Schultz GS, Gibson DJ. A surfactant-based wound dressing can reduce bacterial biofilms in a porcine skin explant model. Int Wound J. 2017 Apr;14(2):408-413. doi: 10.1111/iwj.12619. Epub 2016 May 22. PMID 27212453
- [Background] Salisbury AM, Percival SL. Efficacy of a Surfactant-Based Wound Dressing in the Prevention of Biofilms. Adv Skin Wound Care. 2018 Nov;31(11):514-520. doi: 10.1097/01.ASW.0000544612.28804.34. PMID 30335643
- [Background] Mayer D, Armstrong D, Schultz G, Percival S, Malone M, Romanelli M, Keast D, Jeffery S. Cell salvage in acute and chronic wounds: a potential treatment strategy. Experimental data and early clinical results. J Wound Care. 2018 Sep 2;27(9):594-605. doi: 10.12968/jowc.2018.27.9.594. PMID 30204575
- [Background] Pittinger TP, Curran D, Hermans MH. The treatment of paediatric burns with concentrated surfactant gel technology: a case series. J Wound Care. 2020 Jun 1;29(Sup6):S12-S17. doi: 10.12968/jowc.2020.29.Sup6.S12. PMID 32530755
- [Background] Pittinger T, Curran D, Hermans M. Treatment of Burns in Adult Patients With a Concentrated Surfactant Gel: A Real-life Retrospective Evaluation. Wounds. 2020 Dec;32(12):339-344. PMID 33472159
- [Background] Kirsner RS, Amaya R, Bass K, Boyar V, Ciprandi G, Glat PM, Percival SL, Romanelli M, Pittinger TP. Effects of a surfactant-based gel on acute and chronic paediatric wounds: a panel discussion and case series. J Wound Care. 2019 Jun 2;28(6):398-408. doi: 10.12968/jowc.2019.28.6.398. PMID 31166855